CLINICAL TRIAL: NCT00941395
Title: Enhanced Smoking Cessation for University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-0351; NCI-2018-02552 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0351 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); R01CA069425 (NIH)
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Cigarette Smoker; Current Every Day Smoker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (smoker, survey) (Experimental): Participants who currently smoke complete a survey over 30 minutes and discuss the survey results with the counselor over 30 minutes at week 2. Participants also complete 3 internet surveys over 20 minutes.
  Interventions: Other: Survey Administration
- Arm II (non-smoker, survey) (Experimental): Participants who currently do not smoke complete a survey over 30 minutes and discuss the survey results with the counselor over 30 minutes at week 2.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete surveys

SUMMARY:
This trial studies how well a new smoking cessation and prevention intervention works in enhancing smoking cessation for university students. The new intervention may be easier to use for students to quit smoke.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the feasibility of a new smoking cessation and prevention intervention including two new modules addressing alcohol use and depression.

II. Demonstrate the feasibility of a smoking prevention website.

OUTLINE: Participants are assigned to 1 of 2 arms.

ARM I: Participants who currently smoke complete a survey over 30 minutes and discuss the survey results with the counselor over 30 minutes at week 2. Participants also complete 3 internet surveys over 20 minutes.

ARM II: Participants who currently do not smoke complete a survey over 30 minutes and discuss the survey results with the counselor over 30 minutes at week 2.

After completion of study, participants are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* CESSATION ARM: Student at University of Houston Central Campus or Texas A&M University
* CESSATION ARM: Smoke 1 or more cigarettes a day
* CESSATION ARM: Speak and read English
* CESSATION ARM: Signed informed consent and an acknowledgement of participation requirements
* CESSATION ARM: Be enrolled in at least one class at respective campus at baseline
* CESSATION ARM: Provide current contact information
* CESSATION ARM: Have access to the Internet
* PREVENTION ARM: Student at University of Houston Central Campus or Texas A&M University
* PREVENTION ARM: Speak and read English
* PREVENTION ARM: Signed Informed Consent and an acknowledgement of participation requirements
* PREVENTION ARM: Be enrolled in at least one class at respective campus at baseline
* PREVENTION ARM: Provide current contact information
* PREVENTION ARM: Have access to the Internet
* PREVENTION ARM: Evidence of smoking susceptibility (as defined by the Smoking Susceptibility Scale)
* CESSATION ARM: Willing to answer all survey questions on all survey instruments throughout the duration of study
* PREVENTION ARM: Willing to answer all survey questions on all survey instruments throughout the duration of study

Exclusion Criteria:

* CESSATION ARM: Evidence of major depressive disorder (as defined by PHQ-9 [Patient Health Questionnaire-9])
* CESSATION ARM: Evidence of severe alcohol abuse (as defined by AUDIT [Alcohol Use Disorders Identification Test] measure)
* PREVENTION ARM: Current tobacco use
* PREVENTION ARM: Does not plan to continue as a student at their campus for at least one more year
* CESSATION ARM: Does not plan to continue as a student at their campus for at least one more year
* PREVENTION ARM: Evidence of major depressive disorder (as defined by PHQ-9 [Patient Health Questionnaire-9])
* PREVENTION ARM: Evidence of severe alcohol abuse (as defined by AUDIT measure)
* CESSATION ARM: Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-06-30 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
The ease of use and appeal of various features of the program | Up to 5 months
The quality of the interactive multi-media presentations and their ability to generate interest in smoking cessation and prevention | Up to 5 months
Behavior modification determined by EVOLVE Follow up Survey-Smoker | Up to 5 months
Knowledge of modules in the program | Up to 5 months
Feasibility defined as 90% of the student participants indicating that the intervention program is easy to use and can fit into their schedule | Up to 5 months
  Associations between the dependent variables and smoking status will be evaluated with linear and logistic regression models with campus of origin and smoking status as independent predictors of these outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Prokhorov, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Texas A&M, College Station, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org